CLINICAL TRIAL: NCT06997393
Title: Prevention of Hand Eczema Among Workers in the Fishing Industry in Greenland: an Intervention Study
Brief Title: Prevention of Hand Eczema Among Workers in the Fishing Industry in Greenland
Acronym: HEFIG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: LEO Foundation (Unknown); University of Copenhagen (Other); Greenland University (Unknown); Government of Greenland, Agency for Health and Prevention (Unknown)
Responsible Party: Principal Investigator, Mathilde Tuborg Andersen, MD, Principal Investigator, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LF-ST-24-500016; 2024-15101 (Other: Science Ethics Committee in Greenland)
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hand Eczema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention programme (Experimental): The participants will have access to a prevention programme.
  Interventions: Behavioral: Prevention programme
- Control group (No Intervention): The participants will not have access to a prevention programme.

INTERVENTIONS:
Behavioral: Prevention programme — The prevention programme consists of a validated educational video and training in the basic recognition and prevention of hand eczema.
  Arms: Prevention programme

SUMMARY:
This study aims to investigate the effect of a prevention programme on hand eczema among workers in the Greenlandic fishing industry. This is a non-randomised clinical trial including employees at four of Royal Greenland's fish processing facilities in Greenland.

ELIGIBILITY:
Inclusion Criteria:

* Employee in Royal Greenland, a state-owned company and one of the largest seafood enterprises in the world
* Written informed consent

Exclusion Criteria:

* Age below 18 years
* Inability to understand the Greenlandic, Danish or English language
* Pregnancy
* Other chronic skin diseases on the hands
* Receiving immunomodulatory therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in knowledge of hand eczema at 3 months | From enrollment to the end of intervention at 12 weeks
  Knowledge of hand eczema measured by a self-reported questionnaire
Change from baseline in clinical severity of hand eczema at 3 months | From enrollment to the end of intervention at 12 weeks
  Clinical severity of hand eczema measured by Hand Eczema Severity Index (HECSI). The HECSI score ranges from 0 to 360, with higher scores reflecting greater disease severity.

SECONDARY OUTCOMES:
Change from baseline in patient-reported quality of life at 3 months | From enrollment to the end of intervention at 12 weeks
  Patient-reported quality of life measured by Hand Eczema Impact Scale (HEIS). The HEIS is a validated 9-item questionnaire that measure the impact of hand eczema on patients' quality of life, based on recall over the past week. Domains include proximal daily activity limitations, embarrassment with the appearance of the hands, frustration with chronic hand eczema, sleep, work, and physical functioning. Each item is scored on a 5-point scale ranging from 0 (not at all) to 4 (extremely). The HEIS score is the average of the 9 items.
Change from baseline in Patient Global Assessment of Disease Severity (PaGA) at 3 months | From enrollment to the end of intervention at 12 weeks
  The PaGA rates the severity of the patient's global disease assessed by the patient and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Change from baseline in the number of self-reported days with absence from work due to hand eczema at 3 months | From enrollment to the end of intervention at 12 weeks
  The number of self-reported days with absence from work due to hand eczema measured by a questionnaire-based interview.
Change from baseline in the number of participants being forced to change their job due to hand eczema at 3 months | From enrollment to the end of intervention at 12 weeks
  The number of participants being forced to change their job due to hand eczema measured by a questionnaire-based interview.
Change from baseline in the availability of protective equipment at 3 months | From enrollment to the end of intervention at 12 weeks
  The availability of protective equipment (protective gloves, cotton undergloves, moisturisers, and disinfectants) at the workplace measured by a questionnaire-based interview.

CONTACTS AND LOCATIONS:
Locations (4):
- Greenland (4):
  - Royal Greenland, Ilulissat
  - Royal Greenland, Maniitsoq
  - Royal Greenland, Qasigiannguit
  - Royal Greenland, Sisimiut

IPD SHARING:
Plan to Share IPD: Undecided